CLINICAL TRIAL: NCT06529237
Title: Plasmodium Falciparum Molecular Surveillance in Mozambique to Monitor Markers of Antimalarial Drug Resistance, Rapid Tests Diagnostic Failure and Transmission in Mozambique: Phase 2
Brief Title: Malaria Molecular Surveillance in Mozambique (Phase 2)
Acronym: GenMoz2
Status: Recruiting | Type: Observational
Sponsor: Centro de Investigacao em Saude de Manhica (Other)
Collaborators: Barcelona Institute for Global Health (Other); University of California, San Francisco (Other); National Malaria Control Program, Mozambique (Unknown)
Responsible Party: Sponsor
Other Study IDs: GenMoz2
Record Dates: First submitted 2024-07-26; First posted 2024-07-31 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Malaria; Falciparum Malaria; Malaria in Pregnancy
Keywords: drug resistance; Diagnostic resistance; Surveillance; Genomics; Importation; Genetic diversity; Plasmodium falciparum; Next Generation Sequencing
MeSH Terms: conditions — Malaria; Malaria, Falciparum

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Dried blood spots on filter paper and rapid diagnostic tests collected by finger-prick
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Children at Health Facilities: Finger-prick sampling (no internvention/clinical trail)
  Interventions: Diagnostic Test: LDH-based malaria rapid diagnostic test
- Pregnant Women at ANC: Finger-prick sampling (no internvention/clinical trail)
  Interventions: Diagnostic Test: Malaria rapid diagnostic test
- All ages: Finger-prick sampling (no internvention/clinical trail)
  Interventions: Diagnostic Test: Malaria rapid diagnostic test

INTERVENTIONS:
Diagnostic Test: LDH-based malaria rapid diagnostic test — Malaria testing using an LDH-based malaria rapid diagnostic test will be added to standard routine testing of suspected cases at health facilities
  Groups: Children at Health Facilities
Diagnostic Test: Malaria rapid diagnostic test — Routine malaria rapid diagnostic tests
  Groups: All ages; Pregnant Women at ANC

SUMMARY:
Mozambique is among the ten countries with the highest burden of malaria worldwide, with an estimated 10.3 million cases in 2021. Malaria transmission is highly heterogeneous across the country, with high burden in the north and very low burden in the south, therefore requiring different strategies for effective control and potential elimination. The GenMoz study (NCT05306067, March 2021-Feb 2024) operationalized a functional malaria molecular surveillance (MMS) system to generate reliable and reproducible temporal genomic data to monitor the effectiveness of rapid diagnostic tests and antimalarials, as well as to continuously characterize transmission levels and sources. The National Malaria Control Program (NMCP) is starting a new strategic cycle (2023-2030) with a plan that includes genomic surveillance for guiding programmatic decisions on six key antimalarial tools : 1. Malaria diagnostics using rapid diagnostic tests (RDTs) based on histidine-rich protein 2 (HRP2); 2. Treatment with artemisinin-based combination therapies (ACTs), including diversification schemes to reduce emergence of resistance; 3. Chemoprevention for pregnant women and children; 4. R21/Matrix-M vaccine rollout; 5. Individual-level interventions in very low transmission settings and 6. Vector control. In Phase 2, the investigators aim to integrate MMS into this wider surveillance framework and scale MMS in Mozambique for quality, timely and appropriate optimization of the public health benefits of the NMCP 2023-2030 strategy in both a proactive and adaptive manner, selecting the combinations of interventions that maximize the impact at the individual and community level.

DETAILED DESCRIPTION:
The AIM of this project is to strengthen and scale Molecular Malaria Surveillance (MMS) in Mozambique for quality, timely, and appropriate optimization of the public health benefits of the NMCP 2023-2030 strategy in both a proactive and adaptive manner, selecting the combinations of interventions that maximize impact at the individual and community level. The SPECIFIC AIMS and expected programmatic impacts are:

AIM 1: Real-time tracking of biological threats to ongoing NMCP strategies:

Address diagnostic failures, including gene deletions in RDT targets (HRP2/3) or non-falciparum infections. Programmatic impacts include updating RDT protocols based on prevalence thresholds of pfhrp2/3 deletions or non-falciparum species.

Assess therapeutic resistance through molecular markers of first-line ACT resistance and support from Therapeutic Efficacy Studies (TES), distinguishing recrudescence from new infections to inform efficacy estimates and containment measures.

Identify transmission sources locally and nationally through genetic case classification and outbreak monitoring, enhancing targeted interventions and source-sink dynamics.

Enhance Anopheles species identification and population structure characterization to improve vector control efficacy through accurate speciation via Vector Molecular Surveillance (VMS).

AIM 2: Develop tools to guide decisions on the value of alternative antimalarial approaches:

Evaluate new chemoprevention methods by assessing resistance markers to preventive antimalarials (SP, AQ, DHAp for IPTp, PMC, SMC, MDA) and model their impact under varying resistance scenarios.

Utilize ANC-based surveillance to inform intervention decisions based on malaria transmission dynamics and monitor ongoing interventions' effectiveness.

Catalog vaccine escape variants to anticipate challenges to vaccine effectiveness post-deployment.

Assess the impact of diversifying ACT regimens on emerging antimalarial resistance through molecular marker analysis.

Conduct parasite genetic diversity surveillance to tailor intervention strategies at a subnational level.

AIM 3: Increase production and uptake of MMS indicators to inform decision-making:

Optimize MMS procedures to maximize the use of GenMoz2 data through improved sampling strategies and digitized data collection tools.

Enhance data sharing and utility for streamlined decision-making via genetic dashboards and integration into NMCP technical group discussions.

Increase NMCP ownership of MMS data through training initiatives and integration into national strategic planning.

Link MMS with broader surveillance systems, clinical trials, and intervention deployments to enhance contextual relevance and effectiveness.

RESULTS-BASED FRAMEWORK

1. Outcomes

   To leverage malaria genomics for optimizing NMCP 2023-2030 strategy, this project will focus on achieving three primary outcomes (PO) and five intermediate outcomes (IO):

   PO 1: Tracking biological threats to ongoing NMCP strategies: Strengthen MMS to detect emerging variants and improve intervention deployment.

   PO 2: Guiding decisions on the value of alternative antimalarial approaches: Develop tools for new MMS applications and create a curated sequence catalog.

   PO 3: Increasing production and uptake of MMS indicators to inform decision-making: Enhance MMS production, sharing, and integration into global health decision-making.
2. Outputs and methodology:

Five workstreams will support these outcomes, facilitating comprehensive malaria control and elimination efforts in Mozambique.

Workstream 1. Sampling In the previous project (GenMoz1), the investigators developed an optimal sampling design for MMS14. For the current project, the investigators will use a multi-cluster probabilistic health facility survey (HFS) to detect pfhrp2/3 deletions and markers of antimalarial resistance, aiming to collect 2840 biological samples. This sampling strategy will be adjusted based on marker prevalence changes over time. The investigators will also conduct dense sampling in districts targeted for elimination and sample pregnant women at their first ANC visit to monitor malaria trends and provide additional biological samples for MMS.

Health facility surveys will involve collecting dried blood spots from 60 RDT-confirmed malaria cases per facility across 10 provinces, aiming to gather high-quality sequence data. For surveillance, a probabilistic approach will be used to select health facilities, focusing on high attendance regions. This will enable us to detect resistance markers with high statistical power.

Targeted sampling will be implement at sentinel health facilities in four districts where therapeutic efficacy studies (TES) are conducted, collecting samples from children with uncomplicated P. falciparum malaria. ANC-based surveillance will monitor malaria at first ANC visits to assess intervention impacts on transmission and help inform public health strategies.

Dense sampling in low-transmission areas will identify transmission sources, monitor outbreaks, and model fine-scale transmission dynamics. Samples will also be collected for vector mosquito surveillance (VMS) to understand Anopheles species diversity and malaria transmission.

Quality control measures include using Redcap tablets for data capture, regular data verification, and systematic sample storage at CISM to maintain DNA integrity. A cascade structure will visually track progress, ensuring data quality and completeness through an internal ShinyDashboard.

Workstream 2. Molecular determinations

Workstream 2 focuses on advanced genomic sequencing techniques to enhance our understanding of malaria parasites and vectors. Multiplexed Amplicon-Based Sequencing (MAD4HatTeR panels) (Output 2.1) aims to sequence 7690 P. falciparum samples, detecting microhaplotypes, pfhrp2/3 deletions, pfcsp polymorphisms, non-falciparum species, and drug resistance markers. A robust bioinformatic pipeline will process data to infer allelic frequencies, identify gene deletions, and standardize data formats. Real-time PCR will complement sequencing by confirming parasite density and genetic variants. CISM will conduct sequencing, with ISGlobal overseeing quality control and providing technical support.

Whole Genome Sequencing (WGS) (Output 2.2) will analyze 500 P. falciparum samples at the Wellcome Sanger Institute to identify genetic markers associated with recrudescence and reinfection, focusing on samples with delayed clearance and treatment failures. Genetic diversity within parasite populations will be assessed using samples collected during health facility surveys in 2022 and 2025, with data shared through MalariaGEN and ENA platforms.

Vector Targeted Sequencing (Output 2.3) will employ the Anospp panel from WSI to study Anopheles species diversity, population structure, and their role in malaria transmission. This high-throughput method enhances vector control efforts by identifying cryptic species and secondary vectors. Collaboration with experts and prioritization of south-south partnerships will explore alternative technologies such as MALDI-TOF MS to improve vector surveillance and control strategies.

Workstream 3. Epidemiological-Genomic Analysis and Modeling

In Workstream 3, the investigators delve into epidemiological-genomic analysis and modeling to enhance our understanding of malaria dynamics and resistance patterns. For Antimalarial Resistance (Output 3.1), the investigators will scrutinize resistance at the provincial level, using bioinformatics pipelines to correct for polyclonality and estimate allele frequencies. Statistical tests will compare resistance marker prevalence across different regions and timeframes, identifying emerging variants of concern. HRP2/3 Deletions (Output 3.2) focuses on assessing pfhrp2/3 deletions using qPCR to validate sequencing methods for detecting gene deletions. TES Outcome Correction (Output 3.3) aims to distinguish between recrudescence and reinfection in therapeutic efficacy studies (TES) using msp1/msp2/polyA genotyping and amplicon sequencing, enhancing evidence for next-generation sequencing-based molecular correction.

In Importation and Transmission (Output 3.4), the investigators will trace malaria transmission and importation sources within provinces through genetic relatedness assessments, incorporating historical data and travel reports. Genetic Diversity Metrics (Output 3.5) involves developing tools to correlate genetic diversity metrics with malaria transmission intensity, informing malaria burden estimates. Vaccine Resistance Monitoring (Output 3.6) focuses on monitoring polymorphisms in the circumsporozoite protein to identify potential vaccine escape variants, providing baseline data for the R21 malaria vaccine's impact. ANC-Based Surveillance (Output 3.7) leverages antenatal care (ANC) data, household-level data, and clinical case reports to model malaria transmission and evaluate intervention impacts, aiding optimal resource allocation.

Malaria Incidence Modeling (Output 3.8) aims to refine malaria incidence estimates by accounting for biases in health-seeking behavior, reporting, and testing, aligning with WHO recommendations. Finally, Modeling Harmonization (Output 3.9) will harmonize modeling activities by integrating genomic and epidemiological data, producing predictive models for malaria transmission and intervention impacts, and guiding malaria control efforts through regular NMCP consultations.

Workstream 4. Data Use

To optimize data utility, genetic data will be integrated into the DHIS2-based iMISS system, enhancing accessibility by combining it with existing case data, entomological surveillance, and intervention data. The iMISS, developed with NMCP collaboration, will be updated with new resistance data and adapted for genetic connectivity and case classification in low transmission areas like Magude district. Formats and visualizations will be defined with stakeholders, with potential use of open-source platforms like Power BI or R Shiny.

Regular semi-annual meetings with NMCP will report on iMISS updates, while MMS and VMS data will be shared in annual regional meetings. Data-driven posters and a quarterly Portuguese brochure will engage healthcare workers and stakeholders. CISM will provide monthly progress reports to NMCP, and advanced training will be offered through workshops and online courses. Annual workshops will build genomics skills, and an MMS contest will incentivize effective sampling.

Integrated surveillance will support initiatives like CHAMPS and serosurveillance of Salmonella Typhi. Capacity building will target NMCP, INS, CISM personnel, and young malaria surveillers. In Mozambique, the NMCP will receive academic and workshop-based training. Angola will benefit from an in-country translational MMS workshop.

INS training will follow a phased approach, starting with qPCR and moving to sequencing. A mentorship period will ensure autonomy in malaria genomics. Quality control will include DBS controls and bioinformatic QC using custom R scripts. VMS capacity building will focus on establishing an NGS-based assay for VMS, with collaboration from vector molecular experts. Three CISM researchers will obtain postgraduate degrees, contributing to MMS capacity, and a specialized module will train students in pathogen surveillance methods.

Workstream 5. Project Management An efficient project management of the project is required to ensure that the activities are conducted timely and with quality. To achieve this, several activities will be conducted. First, a comprehensive operational plan (detailing vendor selection, maintenance schedules, inventory management and transport logistics) will be established to manage procurement, maintenance and logistics to ensure efficient use of resources and minimise delays. Monthly management meetings will monitor financial and resource allocation and a joint tracking document will facilitate these efforts. In addition, a risk mitigation strategy will identify and address potential project risks from the beginning. Second, effective communication and collaboration between stakeholders will be promoted through monthly meetings to provide updates and strategic adjustments, with additional semi-annual meetings with NMCP and regular working group meetings. Programmatic impact will be assessed through policy reviews, meeting minutes, and annual surveys to measure how project-generated evidence informs NMCP malaria control strategies. Third, a monitoring and evaluation (M&E) plan will be developed to ensure timely and comprehensive project tracking. Trimestral assessments will monitor results, with a shared folder for stakeholder access. An annual feedback assessment will facilitate continuous improvement based on stakeholder input. An end-line survey will document lessons learned, identify barriers and facilitators to project success, and inform future strategies. Finally, the project will promote gender equity by highlighting the contributions of Mozambican women scientists through visually appealing posters distributed in educational and public spaces. Activities on the International Day for Women and Girls in Science will highlight the importance of women's participation in science and technology.

ELIGIBILITY:
A) CHILDREN AT HEALTH FACILITIES

Inclusion Criteria:

* Informed, written consent to participate from the guardian
* Children 2-10 years of age
* Fever (axillary temperature ≥37.5ºC) or history of fever in the preceding 24 hours
* At least one positive parasitological test for malaria diagnosis via RDT (HRP2 or LDH)

Exclusion Criteria:

* Unwilling to provide informed, written consent
* Age <2 years or >10 years
* not resident in study area
* Any symptoms of severe malaria
* Negative of both (HRP2 and LDH) parasitological test for malaria via RDT
* History of antimalarial treatment in the last 14 days

B) PREGNANT WOMEN AT ANC

Inclusion Criteria:

* Pregnant women attending first antenatal care visit
* Resident in the study area
* Pregnant Women older than 12 years old
* Informed, written consent to participate from participant and/or guardian

Exclusion Criteria:

* Unwilling to provide informed, written consent
* Not resident in study area
* Any symptoms of severe malaria

C) DENSE SAMPLING

Inclusion Criteria:

* People > 6 months of age
* Fever (axillary temperature ≥37.5ºC) or history of fever in the preceding 24 hours
* Positive parasitological test for malaria diagnosis via RDT
* Informed, written consent to participate from participant and/or guardian

Exclusion Criteria:

* Any symptoms of severe malaria
* Negative parasitological test for malaria via RDT
* Unwilling to provide informed, written consent
* History of antimalarial treatment in the last 14 days

Min Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 1. Children at Health Facilities:
     The first study group comprises children aged 2-10 years who present at health facilities with symptoms suggestive of malaria.
  2. Pregnant Women at Antenatal Care (ANC) Visits:
     The second group includes pregnant women attending their first ANC visit.
  3. General Population for Dense Sampling:
  The third study group involves a diverse population sample of individuals older than 6 months.
Sampling Method: Probability Sample
Enrollment: 18750 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of molecular markers of antimalarial resistance at provincial level | Year 3
Prevalence of hrp2/3 deletions determined at regional level | Year 3
Genetic diversity of the parasite population by period, study area and population | Year 3
Genetic relatedness between pairs of samples and populations by period, study area and population | Year 3
Genetic diversity in circumsporozoite protein C-terminal region encompassing T-cell epitopes | Year 3

CONTACTS AND LOCATIONS:
Locations (1):
- Centro de Investigaçao em Saúde de Manhiça, Manhiça, Maputo Province, Mozambique

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] da Silva C, Matambisso G, Boene S, Rovira-Vallbona E, Pujol A, Comiche K, Sanchez A, Greenhouse B, Chidimatembue A, Aranda-Diaz A, Arnaldo P, Ariani C, Walker P, Mbeve H, Ndimande N, Tembisse D, Ruybal-Pesantez S, Verity R, Rafael B, Candrinho B, Mayor A. Plasmodium falciparum molecular surveillance to inform the Mozambican National Malaria Control Programme strategy: protocol. BMJ Open. 2024 Nov 24;14(11):e092590. doi: 10.1136/bmjopen-2024-092590. PMID 39581722